CLINICAL TRIAL: NCT01258530
Title: A Randomized, Open-label, Single-Dose, Two-Period, Crossover Study to Evaluate the Bioequivalence of Over-encapsulated Oseltamivir Capsules to Marketed Oseltamivir Capsules in Healthy Volunteers
Brief Title: A Study to Evaluate the Bioequivalence of Over-encapsulated Oseltamivir Capsules to Marketed Oseltamivir Capsules in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 115096
Record Dates: First submitted 2010-12-02; First posted 2010-12-13 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Influenza, Human
Keywords: influenza, bioequivalence, oseltamivir, Tamiflu, over-encapsulation
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A (Experimental): Over-encapsulated oseltamivir 75 mg (1 capsule)
  Interventions: Drug: over-encapsulated oseltamivir
- Treatment B (Experimental): oseltamivir 75 mg (1 capsule)
  Interventions: Drug: oseltamivir

INTERVENTIONS:
Drug: over-encapsulated oseltamivir — 75 mg once
  Arms: Treatment A
Drug: oseltamivir — 75 mg once
  Arms: Treatment B

SUMMARY:
This is a study in healthy adult volunteers to assess the bioequivalence of over-encapsulated oseltamivir capsules to commercially available oseltamivir capsules. Both formulations will be administered in the fasting state.

ELIGIBILITY:
Inclusion Criteria:

* AST, ALT, alkaline phosphatase and bilirubin greater than or equal to 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of: Child-bearing potential and agrees to use one of the contraception methods listed in the protocol for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until the follow-up visit.
* Body weight greater than or equal to 50 kg and BMI within the range 18.5 - 31.0 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 ml) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Urinary cotinine levels indicative of smoking or history of regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy, peptic ulceration, inflammatory bowel disease or pancreatitis should be excluded.
* The subject's systolic blood pressure is outside the range of 90-140 mmHg, or diastolic blood pressure is outside the range of 45-90 mmHg or heart rate is outside the range of 50-100 bpm for female subjects or 45-100 bpm for male subjects.
* Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination): Heart rate Males <45 and >100 bpm Females <50 and >100 bpm; PR Interval <120 and >220 msec; QRS duration <70 and >120 msec; QTc interval (Bazett) >450 msec.

Evidence of previous myocardial infarction (Does not include ST segment changes associated with repolarization).

Any conduction abnormality (including but not specific to left or right complete bundle branch block, AV block [2nd degree or higher], Wolf Parkinson White [WPW] syndrome, non-sustained or sustained ventricular tachycardia (greater than or equal to 3 consecutive ventricular ectopic beats).sinus pauses > 3 seconds, or other significant arrhythmia which, in the opinion of the principal investigator and GSK medical monitor, will interfere with the safety of the individual subject.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-12-20 (Actual); Primary Completion 2011-02-03 (Actual); Study Completion 2011-02-03 (Actual)

PRIMARY OUTCOMES:
Plasma oseltamivir carboxylate area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC(0-infinity)) | 9 days
Plasma oseltamivir carboxylate maximum observed concentration (Cmax) | 9 days

SECONDARY OUTCOMES:
Plasma oseltamivir carboxylate area under the concentration-time curve from time zero (pre-dose) to the time of the last quantifiable concentration (AUC(0-t)) | 9 days
Plasma oseltamivir carboxylate terminal phase half-life (t1/2) | 9 days
Plasma oseltamivir carboxylate time of occurrence of Cmax (tmax) | 9 days
Plasma oseltamivir AUC (0-infinity) | 9 days
Plasma oseltamivir AUC(0-t) | 9 days
Plasma oseltamivir Cmax | 9 days
Plasma oseltamivir t1/2 | 9 days
Plasma oseltamivir lag time before observation of drug concentrations in sampled matrix (tlag) | 9 days
Plasma oseltamivir tmax | 9 days
Safety and tolerability of all treatments, including number of subjects with adverse events assessment | 4 weeks
Safety and tolerability of all treatments, including number of subjects with concurrent medications | 4 weeks
Safety and tolerability of all treatments, change from baseline and number subjects with abnormal clinical safety laboratory data | 4 weeks
Safety and tolerability of all treatments, including change from baseline and number of subjects with abnormal ECG assessments | 4 weeks
Safety and tolerability of all treatments, including change from baseline and number of subjects with abnormal vital signs (blood pressure and heart rate) assessments | 4 weeks
Plasma oseltamivir carboxylate lag time before observation of drug concentrations in sampled matrix(tlag) | 9 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 115096 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/115096?search=study&search_terms=115096#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 115096 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115096 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115096 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115096 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115096 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115096 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115096 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register